CLINICAL TRIAL: NCT07041294
Title: 7 mm Versus 5 mm Diameter Immediate Post-Extractive Implants in the Molar Region: A Multicentre Randomised Controlled Trial
Brief Title: Comparing 7 mm and 5 mm Implants Placed Immediately After Molar Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Esposito (Network)
Responsible Party: Sponsor-Investigator, Marco Esposito, Associate Professor, Marco Esposito
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NR430PROT
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Partial Edentulism in the Maxilla or in the Mandible; Immediate Implant Placement
Keywords: Deantal implant; Immediate implant; Post-extraction implant; Wide diameter implant; Follow-up

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician performing the data analysis is masked to the treatment allocation in order to prevent bias during statistical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7 mm Diameter Implant (Experimental): Participants receive a 7 mm diameter implant placed immediately after molar extraction.
  Interventions: Device: 7 mm Diameter Dental Implant
- 5 mm Diameter Implant (Active Comparator): Participants receive a 5 mm diameter implant placed immediately after molar extraction.
  Interventions: Device: 5 mm Diameter Dental Implant

INTERVENTIONS:
Device: 7 mm Diameter Dental Implant — To evaluate immediate post-extraction implants with different diameters (7 vs. 5 mm)
  Arms: 7 mm Diameter Implant
Device: 5 mm Diameter Dental Implant — To evaluate immediate post-extraction implants with different diameters (5 vs. 7 mm)
  Arms: 5 mm Diameter Implant

SUMMARY:
This clinical study aims to evaluate the performance and long-term outcomes of immediate dental implants placed in molar sites after tooth extraction. Eligible patients will receive one implant and a single crown in a posterior area (first or second molar). The study will compare implant and crown success over a five-year period, tracking complications, bone changes, aesthetics, and patient satisfaction. Participants must be at least 18 years old and have sufficient bone to allow immediate implant placement. This research will provide important data on the safety and reliability of immediate implants in posterior areas.

DETAILED DESCRIPTION:
This multicentre randomised controlled trial aims to compare the clinical outcomes of 7 mm versus 5 mm diameter dental implants placed immediately after tooth extraction in the molar region. The goal is to assess whether wider diameter implants offer any advantages in terms of implant survival, complications, bone preservation, and patient satisfaction, when placed in fresh extraction sockets.

A total of 70 patients requiring molar tooth extraction and immediate implant placement will be enrolled across 7 centers. Each participant will receive either a 5 mm or a 7 mm diameter implant, allocated randomly. Standardised surgical and prosthetic protocols will be followed.

Follow-up visits will assess implant stability, radiographic bone changes, and clinical outcomes over time. Patient-reported outcomes and complications will also be recorded to compare the two groups. Results will be reported at 1 and 5 years after loading.

This study may help clinicians make evidence-based decisions when choosing the diameter of implants in molar regions, particularly in immediate post-extraction situations.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to sign an informed consent form
* requiring at least one immediate post-extractive implant in first and/or second molar sites
* sufficient bone to allow placement of an immediate implant at least 7 mm in length and 7 mm in diameter

Exclusion Criteria:

* general contraindications to implant surgery
* immunosuppressed or immunocompromised
* irradiation in the head or neck area
* uncontrolled diabetes
* pregnancy or lactation
* untreated periodontitis
* poor oral hygiene and motivation
* addiction to alcohol or drugs
* psychiatric disorders
* unrealistic expectations
* acute infection (abscess) in the site intended for implant placement
* necessity to lift the maxillary sinus epithelium
* unable to commit to 5-year follow-up post-loading
* under treatment or had previous treatment with intravenous amino-bisphosphonates
* lack of bony wall completely surrounding the future implant
* participation in other studies interfering with present protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of failed crowns (not placed or remade due to implant/prosthetic failure) | From implant placement to 5 years after loading.
  whether it will not be possible to place the crown because of implant failure or secondary to implant failure, or crown that has to be remade for any reason.
Number of failed implants (implant mobility, infection, or mechanical complications) | From implant placement to 5 years post loading.
  Implant failure is defined as implant mobility and/or any infection dictating implant removal, and or/any mechanical problems rendering the implant unusable. The stability of each individual implant will be measured by the independent and blinded outcome assessor manually with a reverse torque of 20 Ncm at abutment connection and at delivery of the definitive crown, or by assessing the stability of the crown, using the handles of two metallic instruments, at 1 and 5 years after loading.
Biological and biomechanical complications | From implant placement to 5 years after loading.
  Biological and biomechanical complications will be recorded and reported by study group. Examples of biological complications are: fistula, peri-implantitis. Examples of biomechanical complications are fracture of the metal screws, loosening of the crown, fracture of ceramic.

SECONDARY OUTCOMES:
Peri-implant marginal bone level changes | From implant placement to 5 years after loading.
  Digital intraoral periapical radiographs will be made with the paralleling technique at implant placement, implant loading, 1 and 5 years after loading. In case of unreadable radiograph, the radiograph has to be made again. Radiographs will be converted to TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known implant length or the diameter of the implant collar. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured at both mesial and distal sides and averaged. Bone level at single implants will b
Aesthetic evaluation | From implant placement to 5 years after loading.
  Aesthetic evaluation of the clinical pictures, taken at delivery of the final restorations, 1 and 5 years follow-ups, on a computer screen by an independent blinded dentist. The pictures of the vestibular and occlusal aspects have to include the 2 adjacent teeth, when present. The aesthetic evaluation will be done following the pink aesthetic score(1).
Patient satisfaction | From implant placement to 5 years after loading.
  At the delivery of the final restorations, 1 and 5 years follow-up the independent outcome assessor at each centre will ask to the patient the following questions:
  1. Are you satisfied with the function of your implant supported tooth? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2. Are you satisfied with the aesthetic outcome of your implant supported tooth? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3. Would you undergo the same therapy again? Possible answers: "yes" or "no".

CONTACTS AND LOCATIONS:
Overall Officials: Marco Esposito, Dentistry, Principal Investigator — IRCCS San Raffaele Scientific Institute and Vita-Salute San Raffaele University, Milan, Italy
Locations (1):
- Nobel dental clinic, Tirana, Albania

REFERENCES:
- [Result] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569

DOCUMENTS (1):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT07041294/Prot_000.pdf